CLINICAL TRIAL: NCT01188928
Title: A Phase 3 Study Comparing Once Daily Treatment With Calcipotriol 50 mcg/g Plus Betamethasone 0.5 mg/g (as Dipropionate) Topical Suspension With Betamethasone 0.5 mg/g (as Dipropionate) in the Topical Suspension Vehicle, Calcipotriol 50 mcg/g in the Topical Suspension Vehicle and the Topical Suspension Vehicle Alone in Subjects With Psoriasis Vulgaris on Non-scalp Regions of the Body (Trunk and/or Limbs)
Brief Title: LEO 80185 in the Treatment of Psoriasis Vulgaris on the Non-scalp Regions of the Body (Trunk and/or Limbs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 80185-G23
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2016-12

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Betamethasone; betamethasone-17,21-dipropionate; Suspensions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 80185 (Experimental): Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) topical suspension
  Interventions: Drug: Calcipotriol plus betamethasone
- Betamethasone (Active Comparator): Betamethasone 0.5 mg/g (as dipropionate) in the topical suspension vehicle
  Interventions: Drug: Betamethasone-17,21-dipropionate
- Calcipotriol (Active Comparator): Calcipotriol 50 mcg/g in the topical suspension vehicle
  Interventions: Drug: Calcipotriene
- Topical suspension vehicle (Placebo Comparator): The topical suspension vehicle alone
  Interventions: Drug: Topical suspension vehicle

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone — Topical suspension once daily for up to 8 weeks.
  Arms: LEO 80185
Drug: Betamethasone-17,21-dipropionate — Topical suspension once daily for up to 8 weeks.
  Arms: Betamethasone
Drug: Calcipotriene — Topical suspension once daily for up to 8 weeks.
  Arms: Calcipotriol
Drug: Topical suspension vehicle — Topical suspension once daily for up to 8 weeks.
  Arms: Topical suspension vehicle

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Calcipotriol 50 Mcg/g Plus Betamethasone 0.5 mg/g (as Dipropionate) Topical Suspension with the active components when used individually as monotherapy in the topical suspension vehicle (betamethasone dipropionate in the topical suspension vehicle, calcipotriol in the topical suspension vehicle) and with the topical suspension vehicle alone in the treatment of psoriasis vulgaris on the non-scalp regions of the body (trunk and/or limbs) in a large phase 3 study. This comparison will ensure a more informed assessment of the benefit/risk ratio of Calcipotriol 50 Mcg/g Plus Betamethasone 0.5 mg/g (as Dipropionate) Topical Suspension while also establishing the optimal treatment duration in psoriasis vulgaris on the non-scalp regions of the body (trunk and/or limbs).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained prior to any trial related activities (including any washout period).
* Aged 18 years or above
* Either sex
* Any race or ethnicity
* Attending a hospital outpatient clinic or the private practice of a board certified dermatologist.
* Clinical diagnosis of stable plaque psoriasis vulgaris of at least 6 months duration involving the non-scalp regions of the body (trunk and/or limbs) amenable to treatment with a maximum of 100 g of topical medication per week.
* An investigator's global assessment of disease severity (IGA) of mild or moderate on the body (trunk and/or limbs) at Day 0 (Visit 1).
* A minimum modified Psoriasis Area and Severity Index (PASI) score for extent of 2 in at least one body region (i.e. psoriasis affecting at least 10% of arms, and/or 10% of trunk, and/or 10% of legs)
* Females of childbearing potential must have a negative pregnancy test at Day 0 (Visit 1).
* Females of childbearing potential must agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year) such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomised partner. The patients must have used the contraceptive method continually for at least 1 month prior to the pregnancy test, and must continue using the contraceptive method for at least 1 week after the last application of study medication. A female is defined as not of child-bearing potential if she is postmenopausal (12 months with no menses without an alternative medical cause), or surgically sterile (tubal ligation/section, hysterectomy or bilateral ovariectomy).
* Able to communicate with the investigator and understand and comply with the requirements of the study.

Exclusion Criteria:

* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * etanercept - within 4 weeks prior to randomisation
  * adalimumab, alefacept, infliximab - within 2 months prior to randomisation
  * ustekinumab - within 4 months prior to randomisation
  * experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to randomisation
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, cyclosporine and other immunosuppressants) within 4 weeks prior to randomisation.
* PUVA or Grenz ray therapy within 4 weeks prior to randomisation.
* UVB therapy within 2 weeks prior to randomisation.
* Any topical treatment of the trunk and/or limbs (except for emollients) within 2 weeks prior to randomisation.
* Topical treatment for other relevant skin disorders on the face and flexures (e.g., facial and flexural psoriasis, eczema) with class 1- 5 corticosteroids or vitamin D analogues within 2 weeks prior to randomisation.
* Topical treatment for other relevant skin disorders on the scalp (e.g. scalp psoriasis) with class 1-5 corticosteroids, vitamin D analogues or prescription shampoos within 2 weeks prior to randomisation.
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g. beta blockers, anti-malarials, lithium, ACE inhibitors) during the study.
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
* Subjects with any of the following conditions present on the treatment area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, icthyosis, acne rosacea, ulcers and wounds.
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia.
* Known or suspected severe renal insufficiency or severe hepatic disorders.
* Known or suspected hypersensitivity to component(s) of the investigational products.
* Current participation in any other interventional clinical study.
* Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the 4-week period prior to randomisation or longer, if the class of substance required a longer washout as defined above (e.g. biological treatments).
* Planned excessive exposure to the sun during the study that may affect the psoriasis vulgaris.
* Previously randomised in this study.
* Females who are pregnant, have a positive pregnancy test at Day 0 (Visit 1), or are breast-feeding. Females of child-bearing potential wishing to become pregnant during the study, or not using an adequate method of contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Menter, MD, Principal Investigator — Division of Dermatology, Baylor Research Institute, USA; Stephen Tyring, MD PhD, Principal Investigator — Center for Clinical Studies; Steven A Davis, MD, Principal Investigator — Dermatology Clinical Research Center of San Antonio; David J Cohen, MD, Principal Investigator — Dermatologic Surgery Specialists; Mark Lee, MD, Principal Investigator — Progressive Clinical Research; Tiffani K Hamilton, MD, Principal Investigator — Atlanta Dermatology, Vein & Research Center; Daniel M Stewart, DO, Principal Investigator — Michigan Center for Research Corp.; John J Goodman, MD, Principal Investigator — Palm Beach Research Center; Terry Jones, MD, Principal Investigator — J&S Studies, Inc; Dow Stough, MD, Principal Investigator — Burke Pharmaceutical Research; Jerry Bagel, MD, Principal Investigator — Psoriasis Treatment Center of Central NJ; James A Solomon, MD PhD, Principal Investigator — Ameriderm Research; George J Murakawa, MD PhD, Principal Investigator — Somerset Skin Centre; Michael Bukhalo, MD, Principal Investigator — Altman Dermatology Associates; Jeffrey Moore, MD, Principal Investigator — Deaconess Clinic, Inc.; Jaime D Weisman, MD, Principal Investigator — Peachtree Dermatology Associates Research Center; Jonathan Kantor, MD, Principal Investigator — North Florida Dermatology Associates; David Rodriguez, MD, Principal Investigator — Dermatology Associates and Research; Leonard Swinyer, MD, Principal Investigator — Dermatology Research Center, Inc; Alicia Bucko, MD, Principal Investigator — Academic Dermatology Associates; Johnathan Weiss, MD, Principal Investigator — Gwinnett Clinical Research Center, Inc; William P Werschler, MD, Principal Investigator — Premier Clinical Research; Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; James Swinehart, MD, Principal Investigator — Colorado Medical Research Center, Inc.; Steve Kempers, MD, Principal Investigator — Minnesota Clinical Study Center; Dale Martin, MD, Principal Investigator — Skin Surgery Medical Group, Inc.; Scott Guenthner, MD, Principal Investigator — Indiana Clinical Trials Center; Kenneth Dawes, MD, Principal Investigator — Dawes Fretzin Clinical Research Group; Scott Glazer, MD, Principal Investigator — Glazer Dermatology; Karl G Heine, MD, Principal Investigator — Karl G. Heine, M. D. Dermatology; Fasahat Hamzavi, MD, Principal Investigator — Hamzavi Dermatology; Joseph Samady, MD, Principal Investigator — Dermatology Specialists, Inc.; Artis P Truett III, MD, Principal Investigator — Owensboro Dermatology Associates; Phoebe Rich, MD, Principal Investigator — Oregon Dermatology and Research Center; Robin Shecter, DO, Principal Investigator — VISIONS CLINICAL RESEARCH; Robert Haber, MD, Principal Investigator — Haber Dermatology and Cosmetic Surgery; David Kerr, MD, Principal Investigator — Horizons Clinical Research Center, LLC; David Fivenson, MD, Principal Investigator — David Fivenson, MD Dermatology, PLC; Walter Nahm, MD PhD, Principal Investigator — Walter Nahm, MD, Ph.D., Inc; Steven Grekin, DO, Principal Investigator — Grekin Skin Institute; Joseph F Fowler, MD, Principal Investigator — Dermatology Specialists; Jose E Mendez, DO, Principal Investigator — International Dermatology Research, Inc.; David M Stoll, MD, Principal Investigator — Dermatology Research Centers; Paul S Yamauchi, MD, Principal Investigator — Clinical Science Institute; Robert Nossa, MD, Principal Investigator — The Dermatology Group, PC; Chernila Selbert Alan, MD, Principal Investigator — DBA Torrance Clinical Research; Brent M Boyce, MD, Principal Investigator — Great Lakes Research Group, Inc; David B Friedman, MD, Principal Investigator — Advanced Clinical Research Institute; Andrew King, MD, Principal Investigator — King-Maceyko Dermatology Associates; Catherine Hren, MD, Principal Investigator — Triangle Medical Research Associates, LLC; Elyse S Rafal, MD, Principal Investigator — Derm Research Center of New York; John Siebenlist, MD, Principal Investigator — West Dermatolgy; Linda Stein Gold, MD, Principal Investigator — Henry Ford Health System; Laura K Ferris, MD PhD, Principal Investigator — University of Pittsburgh Medical Center; Elizabeth Hughes Tichy, MD, Principal Investigator — Clinical Trials of Texas, Inc.; Jane M Lee, MD, Principal Investigator — Anderson & Collins Clinical Research, Inc.; Charles P Hudson, MD, Principal Investigator — Hudson Dermatology; Amy M Morris, MD, Principal Investigator — Horizon Research Group, Inc.; Lawrence Green, MD, Principal Investigator — Lawrence J. Green, MD, LLC
Locations (59):
- United States (59):
  - Horizon Research Group, Inc, Mobile, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - DBA Torrance Clinical Research, Lomita, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Walter Nahm, MD, Ph.D., Inc, San Diego, California
  - Coastal Medical Research Group, Inc., San Luis Obispo, California
  - Clinical Science Institute, Santa Monica, California
  - Dermatology Research Centers, Santa Monica, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Dermatology Associates and Research, Coral Gables, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia
  - Peachtree Dermatology Associates, Atlanta, Georgia
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - Gwinnett Clinical Research Center, Inc, Snellville, Georgia
  - Altman Dermatology Associates, Arlington Hts, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Hudson Dermatology, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Lawrence J. Green, MD, LLC, Rockville, Maryland
  - David Fivenson, MD Dermatology, PLC, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc, Bay City, Michigan
  - Michigan Center for Research Corp.,, Clinton Township, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Karl G. Heine, M. D. Dermatology, Henderson, Nevada
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - Anderson & Collins Clinical Research, Inc., Edison, New Jersey
  - The Dermatology Group, PC, Verona, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Derm Research Center of New York, Stony Brook, New York
  - Triangle Medical Research Associates, LLC, Cary, North Carolina
  - Haber Dermatology and Cosmetic Surgery, South Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - King-Maceyko Dermatology Associates, Johnstown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - J&S Studies, Inc., College Station, Texas
  - Division of Dermatology, Baylor Research Institute, Dallas, Texas
  - Centre for Clinical Studies, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Progressive Clinical Research, P.A., San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject's first visit was on 27-SEP-2010 and the last subject's last visit was on 29-MAR-2011. Hence the study had a duration of 26 weeks.
Period: Overall Study
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Started | 482 | 479 | 96 | 95
Completed | 444 | 417 | 82 | 77
Not Completed | 38 | 62 | 14 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle | Total
Number analyzed (Participants) | 482 | 479 | 96 | 95 | 1152
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.4) | 48.5 (13.8) | 48 (13.7) | 49.4 (13.0) | 48.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 193 | 36 | 35 | 462
  Male | 284 | 286 | 60 | 60 | 690
Region of Enrollment [Number; unit: participants]
  United States | 482 | 479 | 96 | 95 | 1152

OUTCOME MEASURES:

1. Primary Outcome: Controlled Disease According to the Investigator's Global Assessment of Disease Severity (IGA) at Weeks 4
Description: The IGA was chosen as the primary efficacy assessment. The primary endpoint is subjects with 'Controlled disease' according to the IGA. 'Controlled disease' is defined as clear or almost clear for subjects with moderate disease at baseline and clear for subjects with mild disease at baseline.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Number analyzed (Participants) | 482 | 479 | 96 | 95
participants | 64 | 60 | 5 | 2

2. Primary Outcome: Controlled Disease According to the Investigator's Global Assessment of Disease Severity (IGA) at Weeks 8
Description: as for outcome 1
Time Frame: week 8
Measure: Number; unit: participants
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Number analyzed (Participants) | 482 | 479 | 96 | 95
participants | 140 | 103 | 14 | 6

3. Secondary Outcome: Mean Percentage Change in PASI From Baseline to Week 4
Description: At all treatment phase visits the (sub)investigator made an assessment of the extent and severity of clinical signs of the subject's psoriasis using a modified PASI score (Psoriasis Area and Severity Index) To make up the score, the three features of a psoriatic plaque redness, scaling and thickness are each assigned a number from 0 to 4 with 4 being worst. The extent of involvement of each region of the body is scored from 0 to 6. Adding up the scores give a range of 0 to 72.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in PASI
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Number analyzed (Participants) | 482 | 479 | 96 | 95
percentage of change in PASI | -46.4 (30.2) | -42.7 (29.4) | -32.2 (27.3) | -17.4 (36.8)

4. Secondary Outcome: Mean Percentage Change in PASI From Baseline to Week 8
Description: as for outcome 3
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in PASI
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Number analyzed (Participants) | 482 | 479 | 96 | 95
percentage of change in PASI | -55.8 (34.4) | -48.6 (35.8) | -43.6 (34.1) | -20.9 (49.1)

ADVERSE EVENTS:
Arm/Group | LEO 80185 | Betamethasone | Calcipotriol | Topical Suspension Vehicle
Serious Adverse Events (participants affected / at risk) | 1/482 | 7/479 | 0/96 | 1/95
Other Adverse Events (participants affected / at risk) | 14/482 | 15/479 | 5/96 | 3/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 80185 (N=482) | Betamethasone (N=479) | Calcipotriol (N=96) | Topical Suspension Vehicle (N=95)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80185 (N=482) | Betamethasone (N=479) | Calcipotriol (N=96) | Topical Suspension Vehicle (N=95)
Nasopharyngitis (Infections and infestations) | 14 | 15 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting or presenting a manuscript relating to the clinical trial to a publisher, reviewer, or other outside person, the Investigator shall provide to LEO a copy of all such manuscripts, and LEO shall have rights to review and comment. Upon the request of LEO the Investigator shall remove any confidential information (other than results generated by the Investigator) prior to submitting or presenting the manuscripts.